CLINICAL TRIAL: NCT07257640
Title: The Safety and Efficay Investigation of IL-5 CAR-T Cell Therapy for Patients With Refractory/Relapsed Eosinophilic Leukemia
Brief Title: IL-5 CAR-T Cell Therapy for Refractory/Relapsed Eosinophilic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2025023
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Hematologic Diseases; Neoplasms
Keywords: IL-5 CAR-T; Eosinophil
MeSH Terms: conditions — Hematologic Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells (Experimental): IL-5 CAR-T cells
  Interventions: Drug: IL-5 CAR-T cells

INTERVENTIONS:
Drug: IL-5 CAR-T cells — Each subject receive IL-5 CAR T-cells by intravenous infusion

SUMMARY:
This is an open-label, single-arm clinical study designed to evaluate the efficacy and safety of IL-5 CAR-T cell therapy in the treatment of patients with CD125-positive eosinophilic leukemia.

DETAILED DESCRIPTION:
The IL-5 CAR is composed of full length human IL-5 (hIL-5) fused to the human CD8α hinge and transmembrane domains, followed by the human 4-1BB co-stimulatory domain and the CD3ζ signaling domain. Prior to CAR-T cell infusion, the patients will be subjected to preconditioning treatment. After CAR-T cell infusion, the patients will be evaluated for adverse reactions and efficacy.

The Main research objectives:

To evaluate the safety and efficacy of IL-5 CAR-T cells in patients with CD125-positive eosinophilic leukemia.

The Secondary research objectives:

To investigate the cytokinetic characteristics of IL-5 CAR-T cells in patients with CD125-positive eosinophilic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female patients aged ≥18 years;
* 2.Diagnosis of eosinophilic leukemia (EL) established according to the WHO 2022 diagnostic criteria;
* 3.Interleukin-5 receptor α (IL-5Rα, CD125) is expressed on ≥50% of leukemic blasts.
* 4.Meet any of the following criteria for refractory/relapsed eosinophilic leukemia:
* a) Inadequate response to standard therapy: failure to achieve complete remission (CR) after standard treatments (e.g., imatinib, corticosteroids, interferon-α, chemotherapy, etc.);
* b) Disease progression/relapse within 6 months after achieving remission;
* 5.Serum total bilirubin ≤1.5 × the upper limit of normal (ULN), and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × ULN;
* 6.Left ventricular ejection fraction (LVEF) >50% as assessed by echocardiography;
* 7.Peripheral oxygen saturation (SpO₂) ≥92% on room air (without supplemental oxygen);
* 8.Estimated life expectancy >3 months;
* 9.Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* 10.Women and men of childbearing potential must agree to use appropriate, effective contraception prior to study entry, throughout the study period, and for 6 months after cell infusion (the safety of this therapy for unborn children is unknown and may pose potential risks);
* 11.Patients who are willing to participate in this study and who are able to understand and voluntarily sign the written informed consent form.

Exclusion Criteria:

* 1.History of epilepsy or other central nervous system (CNS) disorders;
* 2.Presence of any of the following:Hepatitis B surface antigen (HBsAg)-positive; Any of HBeAg, HBeAb, or HBcAb positive and detectable hepatitis B virus (HBV) DNA in peripheral blood above the lower limit of detection; Hepatitis C virus (HCV) antibody-positive; Human immunodeficiency virus (HIV) antibody-positive; Positive serologic test for syphilis;
* 3.History of QT interval prolongation or severe cardiac disease;
* 4.Presence of uncontrolled active infection;
* 5.Any condition that, in the opinion of the investigator, may increase the risk to the subject or interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Complete response (CR), and complete response with incomplete hematologic recovery (CRi) | Up to 12 weeks after CAR-T infusion
  The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and PR (partial response).
Duration of remission ,DOR | Up to 1 years after CAR-T infusion
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Overall survival, OS | Up to 1 years after CAR-T infusion
  The time from CAR-T infusion to death due to any cause
Leukemia-Free Survival, LFS | Up to 2 years after Treatment
  The time from CAR-T infusion torecurrence or metastasis

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No